CLINICAL TRIAL: NCT00426946
Title: Phase 3 Reboxetine Treatment in Depressed Children and Adolescents an 8-Week, Open Study
Brief Title: Reboxetine Treatment in Depressed Children and Adolescents an 8-Week, Open Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Geha Mental Health Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACMHC1
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2007-01-25 (Estimated); Status verified 2004-09

CONDITIONS: Depression
Keywords: Depression Children Reboxetine; A diagnosis of major depressive disorder or a dysthimic disorder according to DSM-IV-TR.; Drug naïve or without chronic medication for at least one month.; Only children who agree to participate and whose parents will sign and informed consent form will be included.
MeSH Terms: conditions — Depression | interventions — Reboxetine

INTERVENTIONS:
Drug: Reboxetine

SUMMARY:
The aim of the present study is to prospectively assess the anti-depressant effectiveness of reboxetine in children and adolescents, as compared with fluoxetine, in a randomized controlled open-label trial.

DETAILED DESCRIPTION:
Introduction: Depression is a prevalent disorder involving 3% of children and 8% of adolescents (Birmaher et al, 1996). Reboxetine, a highly selective norepinephrine reuptake inhibitor, is a representative of a fairly new class of antidepressant agents with specificity for the noradrenergic system (Kasper et al., 2000). Long-term clinical trials of reboxetine treatment have demonstrated that reboxetine is significantly more effective than placebo in the treatment of major depression in adult (Versiani et al., 1999) and elderly (> 65 years) (Rampello et al., 2005) patients. These long-term studies demonstrated that rebxetine was well tolerated. Its adverse events were mild in severity and did not require modification of the study medication (Rampello et al., 2005; Versiani et al., 1999). Few reports were published on the use of reboxetine in children and adolescents with attention deficit/hyperactivity disorder (ADHD) (e.g., Mozes et al., 2005). In our previous study (Ratner et al., 2005), we assessed the effectiveness of reboxetine in a 6-week, prospective, open-label study. Thirty-one children and adolescents with ADHD were treated with reboxetine (4 mg/day), with a significant decrease in ADHD symptoms on all scales measured. To the best of our knowledge, no studies were published on the use of reboxetine in the treatment of depressed children.

Fluoxetine is the drug of choice in the treatment of depression in children and adolescents. Fluoxetine was found to be effective and well tolerated in several studies, including double blind controlled ones (e.g., March et al., 2004).

The aim of the present study was to prospectively assess the anti-depressant effectiveness of reboxetine in children and adolescents, as compared with fluoxetine, in a randomized controlled open-label trial.

Methods:

1. The study is a randomized controlled open-label one.
2. Sixty children and adolescents 6-18 years old will participate.
3. Inclusion criteria:

   1. A diagnosis of major depressive disorder or a dysthimic disorder according to DSM-IV-TR.
   2. Drug naïve or without chronic medication for at least one month.
   3. Only children who agree to participate and whose parents will sign and informed consent form will be included.
4. Exclusion criteria:

   1. A diagnosis of a psychotic disorder or bipolar disorder.
   2. Mental retardation.
   3. Alcohol or drug abuse
   4. Chronic medical condition
   5. Girls (> 12 years) will not be included in the study if a possibility of pregnancy during the study exists.
5. All children will undergo a baseline psychiatric assessment by a child and adolescent psychiatrist. In addition, all participants will undergo a physical examination including weight, height, pulse rate and blood pressure, electrocardiogram, blood assessments (blood count, liver and kidney function).
6. After baseline assessment, participants will be included in one of two possible arms:

   1. . An open randomized trial of reboxetine (4 mg per day) vs. fluoxetine (20 mg per day) for 4 weeks. A second psychiatric assessment will then support continuation on the same dosage or an increase to 8 mg reboxetine or 40 mg fluoxetine. All children will be followed and monitored for side effects along the entire study period. If no clinical improvement occurs- the dosage will be gradually decreased. If clinical improvement occurs, the child can continue the treatment according to clinical judgment.
   2. . Children whose low-medium level of depression and lack of suicidality will point to a clinical decision of psychotherapy treatment without drug therapy will undergo a baseline assessment and be assessed again after 4 weeks of psychotherapy. If a decrease in depressive symptoms is noted of less than 40% (CDRS questionnaire) or less than 2 (CGI-I), reboxetine treatment will be initiated (8 week, open label).
7. Rating Scales:

   1. Efficacy scales:

      I. Clinical Global Impression Scale for Depression (CGI-S) (Guy, 1976) II. Clinical Global Impression Improvement (CGI-I (Guy, 1976) III. Children's Depression Inventory CDI (Kovacs, 1985) IV. Children's Depression Rating Scale-Revised (CDRS-R) (Poznanski et al, 1979; Poznanski and Mokros 1996).

      V. Suicide Ideation Questionnaire-Short Version (Reynolds, 1987) VI. Children's Manifest Anxiety Scale (RCMAS) (Reynolds and Richmond, 1985;1997).

      VII. DSM-IV ADHD Scale (DAS) )Spivak et al. 1999)
   2. Measuring autonomic arousal by assessing GSR- galvanic skin response; heart rate variability and EMG. Procompt, Thought Technology Company; Biograph c, Assessment of side effects: I. Weight and height II. Pulse rate and blood pressure III. Electrocardiogram IV. Spontaneous self reports of side effects and assessment of insomnia, somnolence, headache, gastrointestinal complaints, dizziness, agitation and suicidality.

Adverse effects ECG עוררות פיזיולוגית RCMAS SIQ-SV CDRS-R CDI CGI-I CGI-S

* ּ+ + + + + + + T0
* + + + + + T2
* + + + + + + T4
* + T6
* + + + + + + T8
* + + + + + + + T12

T0- Baseline; T2- 2 weeks on reboxetine; T4- 4 weeks on reboxetine; T6- 6 weeks on reboxetine;T8- 8 weeks on reboxetine; T12- 4 weeks after the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of major depressive disorder or a dysthimic disorder according to DSM-IV-TR.
* Drug naïve or without chronic medication for at least one month.
* Only children who agree to participate and whose parents will sign and informed consent form will be included.

Exclusion Criteria:

* A diagnosis of a psychotic disorder or bipolar disorder.
* Mental retardation.
* Alcohol or drug abuse
* Chronic medical condition
* Girls (> 12 years) will not be included in the study if a possibility of pregnancy during the study exists.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2005-01

SECONDARY OUTCOMES:
Children's Depression Inventory CDI (Kovacs, 1985)
Children's Depression Rating Scale-Revised (CDRS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Paz Toren, Principal Investigator — TACMHC
Locations (1):
- Tel Aviv Community Mental Helath Center, Tel Aviv, Israel